CLINICAL TRIAL: NCT00181194
Title: Reducing Asthma Disparities by Improving Provider-Patient Communication About Asthma Severity and Adherence With Therapy
Brief Title: Reducing Asthma Disparities by Improving Provider-Patient Communication
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20021855
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Device: Asthma Control and Communication Instrument

SUMMARY:
The purpose of this study will be to assess the impact of a culturally-sensitive, patient-focused asthma communication instrument (ACCI) designed to enhance provider-patient communication by prompting and guiding providers in assessments of disease severity and discussion of adherence behaviors with minority patients with asthma.

DETAILED DESCRIPTION:
Improving communication between health care providers and their patients is the critical first step in efforts designed to reduce asthma-related health disparities in urban areas. Improving communication will help providers tailor asthma therapies to their patients' needs, and help providers and patients to overcome barriers (e.g., concerns about adverse effects) to adherence with those asthma treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* are able to provide informed consent;
* report physician-diagnosed asthma;
* report asthma symptoms and/or use of short-acting reliever medication at least twice weekly in the past month.

Exclusion Criteria:

* state they do not have asthma;
* have mild intermittent disease
* no recent evidence of disease activity.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2005-05; Primary Completion 2006-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of Provider Assessment of Asthma Severity
Accuracy of Clinician Assessment of Patient Adherence
Assessment of appropriateness of asthma treatment (consistency of care with asthma guidelines
Patient satisfaction with provider-patient communication and medical care

SECONDARY OUTCOMES:
These outcomes include indicators of poor asthma control such as health care service use for asthma exacerbations (unscheduled office visits, ER visits, hospitalizations) and use of oral corticosteroid and overuse of inhaled beta-agonist medications.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory B Diette, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma And Allergy Center, Baltimore, Maryland, United States